CLINICAL TRIAL: NCT06244199
Title: Transition to Cardiac Rehabilitation (T2CR) to Address Barriers of Multimorbidity and Frailty
Acronym: T2CR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IIR 21-177
Record Dates: First submitted 2024-01-26; First posted 2024-02-06 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Cardiovascular Diseases; Cardiac Rehabilitation; Transition of Care
Keywords: cardiovascular diseases; cardiac rehabilitation; transition of care
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: This is a 4-year, 2-site, type 1 hybrid-effectiveness-implementation trial using a randomized controlled design to compare T2CR-facilitated HBCR to Usual Care, an option that can include Promising Practice HBCR (henceforth called "usual HBCR") but without a transition to HBCR.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Key investigators and outcomes assessors at each site will remain blinded to participant group placement. Quantitative study endpoints are assessed by blinded study personnel (i.e., separate from the clinical and study exercise physiologists who treat the patients in the T2CR intervention or usual HBCR).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- T2CR Intervention (Experimental): Participants randomized to the T2CR intervention arm will receive a transitional care program designed to supplement usual care following an acute heart event. Study personnel will follow T2CR Intervention participants for the course of the 12-month study period to assess endpoints in comparison to the Usual Care arm.
  Interventions: Behavioral: T2CR Intervention
- Usual Care (Active Comparator): Participants randomized to the Usual Care are will receive usual care at the discretion of their clinical providers. Study personnel will follow Usual Care participants for the course of the 12-month study period to assess endpoints in comparison to the T2CR intervention arm.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: T2CR Intervention — The T2CR intervention entails two phases. T2CR Phase 1 (Assess and Plan) is a program that occurs during or shortly after hospital discharge that includes completion of a comprehensive risk assessment, development of strategies to address identified risks while restoring function through education regarding living a healthy lifestyle and familiarization and practice of exercise training techniques. T2CR Phase 2 (Implementation and Support) entails a HBCR program that is based on the Promising Practices HBCR but further enriched by insights and strategies developed in T2CR Phase 1 and which also incorporates techniques that maximize the effectiveness and efficiency of exercise training.
  Arms: T2CR Intervention
Other: Usual Care — Participants will receive usual care following an acute heart event that is recommended by their providers, which may include Promising Practices Home-Based Cardiac Rehabilitation (aka Usual HBCR) at both sites or site-based CR at VAPHS.
  Arms: Usual Care

SUMMARY:
Cardiac rehabilitation (CR) is a secondary prevention program for patients with cardiovascular disease (CVD). It is especially valuable as CVD increasingly occurs in combination with comorbidity, frailty, and complexities of care that predispose patients to functional decline, disability, and high costs. Still, few Veterans participate in CR, in part because of the difficult logistics to attend. Promising Practice home-based CR (HBCR) was developed to increase CR participation, but many Veterans remain too limited by comorbidity and frailty for participation. A Transition to CR (T2CR) intervention is a face-to-face program that fosters vital skills, education, insights, motivation, and patient-provider relationships conducive to successful HBCR thereafter. This study compares Veterans eligible for CR who are randomized to T2CR intervention versus usual care. Differences in functional capacity, HBCR participation, and healthy days at home are compared over one year. Patients' experiences and providers' perspectives of barriers and facilitators to T2CR are also compared.

DETAILED DESCRIPTION:
Cardiac rehabilitation (CR) is an evidence-based secondary prevention program for patients with cardiovascular disease (CVD) that aims to stabilize patients clinically and to restore physical function and health after a CVD event. It is well-suited to the needs of the aging Veterans Health Administration's (VHA) aging population which is prone to CVD in a context of comorbidity, frailty, and associated functional decline. Unfortunately, few eligible Veterans participate. Logistic challenges are a key barrier as few VHA site-based CR programs are available. The Promising Practice home-based CR (HBCR) is a VHA initiative that was designed to improve CR participation using a novel home-based approach. While HBCR has been demonstrated to be effective for Veterans who attend, only few participate. Many Veterans eligible for HBCR remain encumbered by comorbidity and frailty, and often lack confidence and/or perceived capacity for home-based formats of care. The Transition to CR (T2CR) intervention is a 2-phase program that aims to improve the process of HBCR and to thereby better respond to Veterans' needs. T2CR Phase 1 is a ~2 day face-to-face program between the initial CVD hospitalization and home that includes comprehensive assessment of holistic risks (CVD and non-CVD), functional limitations, and psychosocial circumstances. Individualized pragmatic plans are formulated to ensure HBCR is feasible, safe, and practical despite aggregate complexity. Goal setting, adherence reinforcements, and education are integrated; exercise practice is emphasized; and consultations for comorbid issues and telemedicine video facilitation are arranged. T2CR Phase 2 is HBCR that is enriched by the orientation, practice, consultations, supports, and goal setting that were initiated in T2CR Phase 1, as well as innovative exercise training techniques for patients who are frail and/or functionally impaired. T2CR is aligned with the already existing Coordinated Transitional Care (C-TraC) Program. C-TraC nurse practitioners currently hone medication management, medical follow-up, and education as hospitalized Veterans transition to home, but do little to guide recovery of physical function. By facilitating referral to the T2CR intervention, C-TraC care will be enhanced. Using a hybrid efficacy-implementation (type 1) design, the Transition to Cardiac Rehabilitation to Address Barriers of Multimorbidity and Frailty study is a randomized controlled trial to study T2CR versus usual HBCR in the VA Pittsburgh and Boston Healthcare Systems. Quantitative endpoints include functional gains (assessed using the Patient Reported Outcomes Measurement Information System [PROMIS] Physical Function measure) over 365 days as well as a 5-Times Sit-To-Stand performance measure. The number of CR sessions attended, rehospitalizations, and Healthy Days at Home will be assessed. Patients' perceptions of feasibility and acceptability of T2CR will also be evaluated. Providers' perceptions of T2CR will be evaluated as well; the Consolidated Framework for Implementation Research (CFIR) framework will be used to structure their insights. Patient and provider feedback will be applied to refine implementation strategies with the goal to ultimately extend T2CR throughout the entire ORH Promising Practices network.

ELIGIBILITY:
Inclusion Criteria:

* Eligible candidates will consist of male and female Veterans hospitalized with:

  * ischemic heart disease (acute myocardial infarction or stable ischemia)
* revascularization (coronary artery bypass grafting or percutaneous coronary intervention)
* valvular heart disease (surgical or percutaneous intervention for mitral regurgitation or aortic stenosis)
* or heart failure (with reduced or preserved ejection fraction)
* All will be recruited while initially hospitalized and must express willingness to consider cardiac rehabilitation as a treatment option, including the possibility of the intervention which could possibly extend the length of their hospitalization (for 2 days maximum).
* Study candidates must also be English speaking and able to provide written informed consent

Exclusion Criteria:

* Veterans with unstable medical condition as indicated by history, physical exam, and/or laboratory findings end-stage disease likely to be fatal within 12 months
* severe cognitive impairment (MiniCog score 0-2)
* history of addictive or behavioral issues that confound safe administration of HBCR
* hearing loss that interferes with participation in the trial
* living in a long-term care living situation prior to the time of hospitalization, no plans to return to independent living after the hospitalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
PROMIS Physical Function SF 10a | 3 months, i.e., baseline to 3-month change
  The Patient Reported Outcomes Measurement Information System (PROMIS) Physical Function V2.0 Short Form 10a is a standardized patient reported index of practical functional capacity. PROMIS physical function instruments measure self-reported capability and functioning of upper extremities (dexterity), lower extremities (walking or mobility), as well as instrumental activities of daily living. The PROMIS Physical Function Short Form 10a is a standardized questionnaire appropriate for comparing large groups. The Physical Function scaled score is applied as the primary outcome at 90 days.

SECONDARY OUTCOMES:
PROMIS Physical Function SF 10a | Baseline to 6-month and 12-month change
  The Patient Reported Outcomes Measurement Information System (PROMIS) Physical Function V2.0 Short Form 10a is a standardized patient reported index of practical functional capacity. PROMIS physical function instruments measure self-reported capability and functioning of upper extremities (dexterity), lower extremities (walking or mobility), as well as instrumental activities of daily living. The PROMIS Physical Function Short Form 10a is a standardized questionnaire appropriate for comparing large groups.
5-Times Sit-to-Stand | Baseline to 3-, 6-, and 12-month change
  The 5-Times Sit-to-Stand is a performance measure of strength and balance that is applied as an index of capacity and disability risk. This is assessed at baseline and 90 days in all participants and to the extent possible, at 180 and 365 days.
Mini-Cog | Baseline to 3-, 6-, and 12-month change
  A brief assessment of cognition which tests visuospatial representation, recall, and executive function. It is scored on a scale of 0-5, with higher scores suggesting better cognitive performance.
Veterans Specific Activity Questionnaire (VSAQ) | Baseline to 3-, 6-, and 12-month change
  Patient reported 13-item assessment of daily activity that estimates functional capacity and also correlates to cardiorespiratory fitness. Scores range from 1-13 metabolic equivalents (METs).
Morley Frailty Scale | Baseline to 3-, 6-, and 12-month change
  The Frail Scale is a 5-item assessment of fatigue, resistance, ambulation, illnesses, and loss of weight. Scores range from 0-5 with a higher number indicating greater frailty.
Cardiac Self-Efficacy Scale | Baseline to 3-, 6-, and 12-month change
  An assessment of a cardiac patient's confidence and coping capacities after a cardiac event. Scored on a scale of 0 to 52, with a higher score indicating higher confidence.
Patient Health Questionnaire 9-item (PHQ-9) | Baseline to 3-, 6-, and 12-month change
  PHQ-9 is a 9 item depression scale. Scores range from 0-27 with a higher score showing the greater possibility of depression.
Pain, Enjoyment, General Activity (PEG) | Baseline to 3-, 6-, and 12-month change
  A 3-item scale to assess pain intensity and interference, and tracking changes in pain over time. The PEG scale includes individual scales in which participants rate their pain level in different areas on a scale of 0-10. The average of the 3 items is the PEG final score, with higher scores representing higher levels of pain.
Rehospitalizations and Emergency Room Visits | 3-months, 6-months, and 12-months
  The number of rehospitalizations and emergency room visits will be assessed at 3-month, 6-month, and 12-month follow-up time points.
Healthy Days at Home | 12-months
  Independent living is assessed as Healthy Days at Home time. This is a summary quality measure that is used for community-living older Veterans, particularly those at higher risk of death of institutionalization.
Cardiac Rehabilitation Participatory Metrics | 3-months, 6-months, 12-months
  Based on established VA Coordinated Transitional Care (C-TraC) metrics, the number of cardiac rehabilitation sessions attended and number of cardiac rehabilitation program completions will be tracked at follow-up time points.
Perception Metrics | 3-months, 6-months, 12-months
  Perceived value of HBCR as a program of education, nutrition, and support versus its value as a program of exercise-training program (each graded 1 [very little] to 5 [very substantial]).
Veterans RAND 12 Item Health Survey (VR-12) | Baseline to 3-, 6-, and 12-month change
  The Veterans RAND 12-Item Health Survey (VR-12) is a standardized questionnaire which evaluates self-reported quality of life. The score is summarized in two parts, a "Physical Health Summary Measure {PCS-physical component score}" and a "Mental Health Summary Measure {MCS-mental component score}." Scoring includes a standardized t-score with a mean of 50 and standard deviation of 10.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel E Forman, MD, Principal Investigator — VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA
Locations (2):
- United States (2):
  - VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts
  - VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No